CLINICAL TRIAL: NCT02393066
Title: A Comparison of Hemodynamic Effects Between Dexmedetomidine and Propofol for Sedation in Patients With Major Abdominal Tumor Surgery
Brief Title: Comparison of Hemodynamics Between Dexmedetomidine and Propofol for Sedation in Patients With Abdominal Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 201407023MINA
Record Dates: First submitted 2014-10-27; First posted 2015-03-19 (Estimated); Last update posted 2015-08-05 (Estimated); Status verified 2015-08

CONDITIONS: Disorder; Mental, Sedative; Pain, Postoperative; Surgery
MeSH Terms: conditions — Pain, Postoperative | interventions — Propofol; Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- propofol (Active Comparator): these patients are sedated with propofol infusion during ICU admission
  Interventions: Drug: Propofol
- dexmedetomidine (Active Comparator): these patients are sedated with dexmedetomidine infusion during ICU admission
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Propofol — Sedation
  Other Names: Propofol-Lipuro
  Arms: propofol
Drug: Dexmedetomidine — Sedation
  Other Names: Precedex
  Arms: dexmedetomidine

SUMMARY:
This is a single-blind randomized clinical trial. Patients undergoing abdominal tumor surgery were recruited to participate in the study. Apart from routine treatment in the surgical intensive care unit, the subjects were randomly divided into two groups: Propofol group (Group P) and Dexmedetomidine group (Group D) and received continuous intravenous infusion of Propofol (infusion dosage range: 0.3 ~ 1.6 mg/kg/h) or Dexmedetomidine (infusion dosage range: 0.1 ~ 0.7 mcg/kg/h) according to their assigned group. Patients' hemodynamic status was monitored using a chest Bioreactance technique, Continuous Non-Invasive Cardiac Output and Hemodynamic Monitor at preset time points (time of recruitment [0h], 2, 4, 6, 12h and 24h). Clinical data such as vital signs, hemodynamic parameters, laboratory results, fluid volume and drugs used were also recorded.

ELIGIBILITY:
Inclusion Criteria:

* non-emergent major abdominal tumor surgery with ICU admission
* the need of sedation during ICU stay

Exclusion Criteria:

* age older than 99 years
* age younger than 20 years
* refractory arrhythmias
* refractory shock status after resuscitation
* new onset of myocardial infarction
* severe heart failure or NYHA 4
* APACHE score > 30 when recruiting
* severe liver cirrhosis or CHILD B or C
* organ transplantation within one year
* pregnancy
* allergic to propofol or dexmedetomidine

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-10; Primary Completion 2015-07 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
cardiac index | six hours after recruitment
  the cardiac index measured by the Bioreactance-based noninvasive CO measurement (NICOM system) six hours after recruitment

SECONDARY OUTCOMES:
mean arterial pressure | six hours after recruitment
heart rate | six hours after recruitment
stroke volume | six hours after recruitment
urine output | six hours after recruitment

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Chang Yeh, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taipei, Taiwan